CLINICAL TRIAL: NCT06206525
Title: Feasibility Trial Using an Insulin Dosing Calculator for Patients With Type 2 Diabetes Mellitus on Hospital Admission
Brief Title: Feasibility Trial Using an Inpatient Insulin Dosing Calculator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Hou-Hsien Chiang, Clinician researcher, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018906; 2T32DK007247-41 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin dosing calculator (Experimental)
  Interventions: Other: Initial insulin dosing using the calculator

INTERVENTIONS:
Other: Initial insulin dosing using the calculator — Participants will receive initial insulin doses by the calculator on hospital admission.

SUMMARY:
The goal of this feasibility trial is to test whether a novel insulin dosing calculator can improve blood glucose management for patients with type 2 diabetes mellitus on hospital admission. The main questions it aims to answer are:

* Whether using this calculator leads to no excessive hypoglycemia?
* Whether using this calculator leads to a decrease of hyperglycemia?

Participants will receive initial insulin doses by the calculator on hospital admission, and the rest of care will follow standard of care. Participants will be compared with patients in the UW observational cohort who received initial insulin doses by standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted to University of Washington Medical Centers
* With history of type 2 and/or steroid-induced diabetes mellitus
* Receiving insulin therapy prior to admission

Exclusion Criteria:

* Patients who are admitted to ICU or obstetrics ward
* Patients who are admitted for elective surgery or procedure
* Patients who present with diabetic ketone acidosis, hyperosmolar hyperglycemic state or require intravenous insulin infusion
* Patients who have no meal intake for 24 hours prior to admission, or planned nothing per oral (NPO) during the first 24 hours after admission
* Patients who report low appetite (25% or less) on admission or have a significantly decreased level of consciousness that they unlikely eat right after admission
* Patients who receive enteral feeding after admission
* Patients who develop severe acute kidney injury needing dialysis therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical significant hypoglycemia | During the first 48 hours after admission
  Participates who develop blood glucose concentration lower than 54 mg/dL

SECONDARY OUTCOMES:
Mean blood glucose concentration (mg/dL) | During the first 24 hours after admission
Clinical significant hyperglycemia | During the first 48 hours after admission
  Participates who develop blood glucose concentration higher or equal to 300 mg/dL
Hypoglycemia lower than 70 mg/dL | During the first 48 hours after admission
  Participates who develop blood glucose concentration lower than 70 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Hou-Hsien Chiang, MD, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Harborview Medical Center, Seattle, Washington
  - UW Medical Center - Northwest, Seattle, Washington
  - UW Medical Center - Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered only on a collaborative basis with PIs, after evaluation of the proposed study protocol and statistical analysis plan.

REFERENCES:
- [Background] Murad MH, Coburn JA, Coto-Yglesias F, Dzyubak S, Hazem A, Lane MA, Prokop LJ, Montori VM. Glycemic control in non-critically ill hospitalized patients: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2012 Jan;97(1):49-58. doi: 10.1210/jc.2011-2100. Epub 2011 Nov 16. PMID 22090269
- [Background] Farrugia Y, Mangion J, Fava MC, Vella C, Gruppetta M. Inpatient hyperglycaemia, and impact on morbidity, mortality and re-hospitalisation rates. Clin Med (Lond). 2022 Jul;22(4):325-331. doi: 10.7861/clinmed.2022-0112. PMID 35882487
- [Background] Bersoux S, Cook CB, Kongable GL, Shu J, Zito DR. Benchmarking glycemic control in u.s. Hospitals. Endocr Pract. 2014 Sep;20(9):876-83. doi: 10.4158/EP13516.OR. PMID 24641927
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Umpierrez GE, Smiley D, Hermayer K, Khan A, Olson DE, Newton C, Jacobs S, Rizzo M, Peng L, Reyes D, Pinzon I, Fereira ME, Hunt V, Gore A, Toyoshima MT, Fonseca VA. Randomized study comparing a Basal-bolus with a basal plus correction insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes: basal plus trial. Diabetes Care. 2013 Aug;36(8):2169-74. doi: 10.2337/dc12-1988. Epub 2013 Feb 22. PMID 23435159
- [Background] Umpierrez GE, Hellman R, Korytkowski MT, Kosiborod M, Maynard GA, Montori VM, Seley JJ, Van den Berghe G; Endocrine Society. Management of hyperglycemia in hospitalized patients in non-critical care setting: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2012 Jan;97(1):16-38. doi: 10.1210/jc.2011-2098. PMID 22223765
- [Background] Chiang HH, Surampudi P, Sood A. Determinants of initial insulin therapy for hospitalized patients with diabetes mellitus. J Diabetes Complications. 2022 Oct;36(10):108307. doi: 10.1016/j.jdiacomp.2022.108307. Epub 2022 Sep 8. PMID 36116360
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 16. Diabetes Care in the Hospital: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S267-S278. doi: 10.2337/dc23-S016. PMID 36507644